CLINICAL TRIAL: NCT02846857
Title: An Open-label, Randomized, Multicenter Study to Assess the Efficacy of Single-hormone Closed-loop Strategy, Dual-hormone Closed-loop Strategy and Sensor-augmented Pump Therapy in Regulating Glucose Levels for 15 Weeks in Free-living Outpatient Conditions in Adolescents and Adults With Type 1 Diabetes
Brief Title: Closed-loop Control of Glucose Levels (Artificial Pancreas) for 15 Weeks in Adolescents and Adults With Type 1 Diabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-17
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Type 1 Diabetes
Keywords: Closed-loop system; Artificial pancreas; Type 1 diabetes; Hypoglycemia; Insulin; Glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance | interventions — Methods; Insulin Infusion Systems; Continuous Glucose Monitoring; Insulin; Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sensor-augmented pump therapy (Active Comparator): Participants will use sensor-augmented pump therapy with low-glucose suspend to regulate glucose levels. The low-glucose suspend feature available in the MiniMed® Paradigm® Veo™, Medtronic combined with the Enlite sensor® will be used. This feature allows for suspension of insulin delivery at a pre-set sensor glucose value for up to 2 hours.
  Interventions: Other: 15-week intervention with sensor-augmented pump; Device: Insulin pump; Device: Continuous glucose monitoring system; Drug: Insulin
- Single-hormone closed-loop strategy (Active Comparator): Variable subcutaneous insulin infusion will be used to regulate glucose levels. Participant's usual fast-acting insulin analog will be infused using a subcutaneous infusion pump (MiniMed® Paradigm® Veo™, Medtronic). Every 10 minutes, the glucose levels as measured by the sensor (Enlite sensor®, Medtronic) will be transferred automatically to a smartphone, that harbors the algorithm, that will calculate the recommended doses and will send it wirelessly to the infusion pump.
  Interventions: Other: 15-week intervention with single-hormone closed-loop; Device: Insulin pump; Device: Continuous glucose monitoring system; Drug: Insulin
- Dual-hormone closed-loop strategy (Active Comparator): Variable subcutaneous insulin and glucagon mini-boluses will be infused using two separate subcutaneous infusion pumps to regulate glucose levels (MiniMed® Paradigm® Veo™, Medtronic). Participant's usual fast-acting insulin analog and Glucagon (Eli Lilly) will be used. Every 10 minutes, the glucose level as measured by the sensor (Enlite sensor®, Medtronic) will be transferred automatically to a smartphone, that harbors the algorithm, that will calculate the recommended doses and will send it wirelessly to the infusion pumps. Newly reconstituted glucagon will be used every 24 hours.
  Interventions: Other: 15-week intervention with dual-hormone closed-loop; Device: Insulin pump; Device: Continuous glucose monitoring system; Drug: Insulin; Drug: Glucagon

INTERVENTIONS:
Other: 15-week intervention with sensor-augmented pump — A sensor will be inserted on the day before the start of the intervention by the participant. The participant will also have to install the study insulin pump. Participants will be advised to continue with study intervention at home for the next 15 weeks. Participants will have been previously shown how to use the study insulin pump.
  Arms: Sensor-augmented pump therapy
Other: 15-week intervention with single-hormone closed-loop — A sensor will be inserted on the day before the start of the intervention by the participant. On the first day of the intervention, participants will be admitted to the clinical research facility anytime between 8:00 am and 11:30 am. Training on connection and disconnection of the system, meal boluses, etc. will be given. Only participants demonstrating competency on use of study devices will be allowed to continue to the home study phase. Participants will be advised to continue with study intervention at home for the next 15 weeks.
  Arms: Single-hormone closed-loop strategy
Other: 15-week intervention with dual-hormone closed-loop — A sensor will be inserted on the day before the start of the intervention by the participant. On the first day of the intervention, participants will be admitted to the clinical research facility anytime between 8:00 am and 11:30 am. Training on connection and disconnection of the system, meal boluses, etc. will be given. Only participants demonstrating competency on use of study devices will be allowed to continue to the home study phase. Participants will be advised to continue with study intervention at home for the next 15 weeks. Participants will have to reconstitute glucagon everyday.
  Arms: Dual-hormone closed-loop strategy
Device: Insulin pump — MiniMed® Paradigm® Veo™, Medtronic
Device: Continuous glucose monitoring system — Enlite sensor®, Medtronic
Drug: Insulin — Participant's usual fast-acting insulin analog will be used: Lispro (Humalog), Aspart (NovoRapid) or Glulisine (Apidra)
Drug: Glucagon — Glucagon (Eli Lilly) will be used during dual-hormone closed-loop strategy.
  Arms: Dual-hormone closed-loop strategy

SUMMARY:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. A dual-hormone closed loop strategy regulates glucose levels through the infusion of two hormones: insulin and glucagon.

The objective of this study is to compare, in a randomized multicenter trial, the effectiveness of single-hormone closed-loop, dual-hormone closed-loop, and sensor-augmented pump therapy with low-glucose suspend in regulating day-and-night glucose levels in outpatient settings for 15 weeks in adolescents and adults.

The investigators hypothesize that dual-hormone closed-loop will reduce time spent in hypoglycemia compared to single-hormone closed-loop, which in turn will be more effective than sensor-augmented pump therapy with low-glucose suspend.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 12 years of old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. The subject will have been on insulin pump therapy for at least 3 months.
4. HbA1c ≤ 11%.

Exclusion Criteria:

1. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
2. Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. History of pheochromocytoma or insulinoma (glucagon could induce a hormonal response of these tumors)
4. Beta-blockers at high dose based on investigator's evaluation of dosage interference with glucagon (glucagon can modify effect of beta-blockers, mostly evident at very high doses)
5. Chronic indometacin treatment (can prevent glucagon effect on liver thus its ability to raise glucose)
6. Chronic acetaminophen treatment (can interfere with glucose sensor measurements)
7. Warfarin chronic treatment if INR monitoring cannot be evaluated (can increase the risk of bleeding)
8. Anticholinergic drug (risk of interaction)
9. Pregnancy.
10. Severe hypoglycemic episode within two weeks of screening.
11. Current use of glucocorticoid medication (except low stable dose and inhaled steroids).
12. Known or suspected allergy to the trial products
13. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
14. Anticipating a significant change in exercise regimen between admissions (i.e. starting or stopping an organized sport).
15. Treatments that could interfere with glucagon

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Percentage of time of glucose levels below 3.9 mmol/L | 15 weeks

SECONDARY OUTCOMES:
HbA1c | 15 weeks
Percentage of time of glucose levels spent in the target range | 15 weeks
  Target range is defined to be between 4 and 10 mmol/L from 7:00 to 22:00 and between 4 and 7.8 mmol/L from 22:00 to 7:00
Area under the curve of glucose levels below 3.9 mmol/L | 15 weeks
Area under the curve of glucose levels below 3.3 mmol/L | 15 weeks
Area under the curve of glucose levels below 2.8 mmol/L | 15 weeks
Percentage of time of glucose levels below 3.3 mmol/L | 15 weeks
Percentage of time of glucose levels below 2.8 mmol/L | 15 weeks
Total number of hypoglycemic events below 3.1 mmol/L | 15 weeks
Percentage of time of glucose levels above 7.8 mmol/L | 15 weeks
Percentage of time of glucose levels above 10.0 mmol/L | 15 weeks
Mean glucose levels | 15 weeks
Standard deviation of glucose levels | 15 weeks
Coefficient of variation of glucose levels | 15 weeks
Total daily dose of insulin | 24 hours
Total daily dose of glucagon | 24 hours
Percentage of time of closed-loop operation | 15 weeks
Percentage of time of glucose sensor availability | 15 weeks
Time between failures due to glucose sensor unavailability | 15 weeks
Time between failures due to pump connectivity | 15 weeks
Percentage of time when patients switched back to insulin pump therapy | 15 weeks
Percentage of time when the closed-loop was automatically switched to insulin pump therapy | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal

IPD SHARING:
Plan to Share IPD: Undecided